CLINICAL TRIAL: NCT01271868
Title: Study of Recombinant Factor IX Product, IB1001, in Previously Treated Pediatric Subjects With Hemophilia B
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medexus Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB1001-02
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia B
Keywords: Recombinant Factor IX
MeSH Terms: conditions — Hemophilia B | interventions — IB1001

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IB1001 (Experimental)
  Interventions: Biological: IB1001

INTERVENTIONS:
Biological: IB1001
  Other Names: Recombinant factor IX; IXINITY

SUMMARY:
The Study's Primary Objective is to evaluate the pharmacokinetics, safety (acute effects associated with infusions, and inhibitor development) and efficacy (breakthrough bleeding and control of hemorrhaging during prophylaxis) of IB1001 in previously treated pediatric subjects with hemophilia B.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent or legal guardian must give written Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent and be willing to make the required study visits and follow instructions while enrolled in the study. For subjects ≥7 years of age, assent will be obtained if required by the institution. For subjects < 7 years of age, legal assent is not reasonable to obtain.
2. Severe (factor IX activity ≤2 IU/dL) hemophilia B subjects currently on-demand therapy with a minimum of 2 bleeding episodes requiring factor IX therapy over the preceding 6 months or 4 bleeding episodes over the preceding 12 months; subjects on prophylaxis with a bleeding pattern similar to that above demonstrated prior to starting prophylaxis
3. Immunocompetent (CD4 count >400/mm3) and not receiving immune modulating or chemotherapeutic agents
4. Previously treated patients with a minimum of 50 exposure days to a factor IX preparation
5. Platelet count at least 150,000/mm3
6. Liver function: alanine transaminase [ALT] and aspartate transaminase [AST] ≤2 times the upper limit of the normal range
7. Total bilirubin ≤1.5 times the upper limit of the normal range
8. Renal function: serum creatinine ≤1.25 times the upper limit of the normal range
9. Willingness to participate in the trial for approximately 6 months (50 exposures)
10. Age ≤12 years
11. Hemoglobin ≥7 g/dL at the time of the blood draw

Exclusion Criteria:

1. History of factor IX inhibitor ≥0.6 Bethesda units (BU)
2. Existence of another coagulation disorder
3. Evidence of thrombotic disease, fibrinolysis, or disseminated intravascular coagulation (DIC)
4. Use of an investigational drug within 30 days prior to study entry
5. On medications that could impact hemostasis, such as aspirin
6. History of poor compliance, a serious medical or social condition, or any other circumstance that, in the opinion of the investigator, would interfere with participation or compliance with the study protocol
7. History of adverse reaction to either plasma-derived factor IX or recombinant factor IX that interfered with the subject's ability to treat bleeding episodes with a factor IX product

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (3):
  - RUSH University Medical Center, Chicago, Illinois
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Gulf States Hemophilia & Thrombophilia Center, Houston, Texas
- India (6):
  - AMRI Hospital, Institute of Haematology & Transfusion Medicine, Kolkata
  - Christian Medical College and Hospital, Ludhiana
  - Jehangir Clinical Development Centre Pvt. Ltd. Jehangir Hospital Premises, Pune
  - Sahyadri Speciality Hospital, Pune
  - Bhailal Amin General Hospital, Vadodara
  - Christian Medical College, Vellore
- Great Ormond Street Hospital for Children, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Pharmacokinetic Study
Arm/Group | IB1001
Started | 9
Completed | 9
Not Completed | 0
Period: Treatment Study
Arm/Group | IB1001
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- IB1001: PK study and Treatment Study
Arm/Group | IB1001
Number analyzed (Participants) | 9
Age, Customized [Number; unit: years]
  0 to 5 years | 3
  6 to 11 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Infusions Required for Bleed Control
Time Frame: Treatment Study: at least 50 ED (approximately 6 months); actual mean subject duration: 39.7 ± 12.4 months
Measure: Count of Units; unit: Number of Infusions
Units Other Than Participants: Number of Infusions
Groups:
- IB1001: Treatment phase: Prophylaxis treatment (n=8) and on demand treatment (n=1)
Arm/Group | IB1001
Number analyzed (Participants) | 9
Number analyzed (Number of Infusions) | 33
Number of Infusions
  0 infusions | 4
  1 infusion | 25
  2 infusions | 1
  3 infusions | 1
  4 infusions | 1
  5 infusions | 1

2. Secondary Outcome: Area Under the Curve (0-inf)
Description: Factor IX levels were assessed at the following time points:
  Pre-infusion, post-infusion at 15-30 min, 4-6 hours, 24-26 hours, 68-72 hours
Time Frame: Pre-infusion to 72 hours following infusion
Population: 9 subjects completed the PK phase. Only 6 subjects had adequate data for formal PK analysis.
Measure: Mean (Standard Deviation); unit: IU*hr/dL
Groups:
- IB1001: PK phase
Arm/Group | IB1001
Number analyzed (Participants) | 6
IU*hr/dL | 1062 (322)

3. Secondary Outcome: Terminal Half-life
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Population: 9 subjects completed the PK phase. Only 6 subjects had adequate data for formal PK analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | IB1001
Number analyzed (Participants) | 6
hours | 22.6 (7)

4. Secondary Outcome: Concentration (Max)
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Population: 9 subjects completed the PK phase. Only 6 subjects had adequate data for formal PK analysis.
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | IB1001
Number analyzed (Participants) | 6
IU/dL | 51.7 (15.7)

5. Secondary Outcome: Incremental Recovery
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Population: 9 subjects completed the PK phase. Only 6 subjects had adequate data for formal PK analysis.
Measure: Mean (Standard Deviation); unit: IU/dL per IU/kg
Arm/Group | IB1001
Number analyzed (Participants) | 6
IU/dL per IU/kg | 0.84 (0.50)

6. Secondary Outcome: Clearance
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Population: 9 subjects completed the PK phase. Only 6 subjects had adequate data for formal PK analysis.
Measure: Mean (Standard Deviation); unit: mL/(kg*hr)
Arm/Group | IB1001
Number analyzed (Participants) | 6
mL/(kg*hr) | 7.3 (3.1)

7. Secondary Outcome: Volume of Distribution (Steady State)
Description: as for outcome 2
Time Frame: Pre-infusion to 72 hours following infusion
Population: 9 subjects completed the PK phase. Only 6 subjects had adequate data for formal PK analysis.
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | IB1001
Number analyzed (Participants) | 6
mL/kg | 244 (166)

8. Secondary Outcome: Annualized Bleed Rate
Description: Measure was assessed during the Treatment Study
Time Frame: Treatment Study: at least 50 ED (approximately 6 months); actual mean subject duration: 41.7+/- 11.7 Months
Measure: Median (Full Range); unit: bleeds/year
Groups:
- IB1001: Treatment study for those receiving prophylaxis treatment (n=8)
Arm/Group | IB1001
Number analyzed (Participants) | 8
bleeds/year | 0.26 [0 to 1.6]

ADVERSE EVENTS:
Groups:
- IB1001: IB1001 Safety population includes all subjects who received at least one dose of IB1001
Arm/Group | IB1001
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IB1001 (N=9)
Vomiting (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 4
Swelling (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Otitis Media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination leading to a small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No